CLINICAL TRIAL: NCT02517749
Title: Randomised Controlled Trial Comparing Outpatient Management of Malignant Pleural Effusion Via an Indwelling Pleural Catheter and Talc Pleurodesis Versus Standard Inpatient Management in Improving Health Related Quality of Life
Brief Title: Out Patient Talc Slurry Via Indwelling Pleural Catheter for Malignant Pleural Effusion Vs Usual Inpatient Management
Acronym: OPTIMUM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: Becton, Dickinson and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RJ115/N175
Record Dates: First submitted 2015-08-05; First posted 2015-08-07 (Estimated); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Pleural Effusion, Malignant
MeSH Terms: conditions — Pleural Effusion, Malignant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care Group (Active Comparator): Patients in this group will be managed as per the British Thoracic Society guideline for management of malignant pleural effusions. They will undergo chest tube insertion and undergo Talc pleurodesis with 4g of SteriTalc
  Interventions: Device: Chest Drain Insertion and Talc Pleurodesis
- Indwelling Pleural Catheter Group (Active Comparator): Patients in this group will undergo Indwelling Pleural Catheter (IPC) insertion. This will be inserted as per standard practice. They will undergo Talc pleurodesis via the IPC with 4g SteriTalc
  Interventions: Device: Indwelling Pleural Catheter Insertion and Talc Pleurodesis

INTERVENTIONS:
Device: Chest Drain Insertion and Talc Pleurodesis
  Arms: Usual Care Group
Device: Indwelling Pleural Catheter Insertion and Talc Pleurodesis
  Arms: Indwelling Pleural Catheter Group

SUMMARY:
This is a multicentre randomised controlled trial evaluating global health related quality of life outcomes in patients with malignant pleural effusions. Patients will be randomised to receive either chest drain and talc pleurodesis or indwelling pleural catheter and talc pleurodesis. Patients will be followed up for 3 months post intervention

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of malignant pleural effusion
2. WHO performance status 2 or less unless performance status is impaired by presence of effusion and likely to significantly improve with drainage
3. Expected survival greater than 3 months

Exclusion Criteria:

1. Age less than 18 years old
2. Pregnant or lactating
3. Known allergy to Talc or Lignocaine
4. Lack of symptomatic relief from effusion drainage
5. At least twice weekly drainage cannot be undertaken
6. Lymphoma or small cell carcinoma except*:

   1. Failure of chemotherapy
   2. Deemed for palliative management
7. Non malignant effusions
8. Loculated pleural effusion
9. Unable to provide written informed consent to trial participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Global health-related quality of life | 30 days
  Global health related quality of life as measured by EORTC QLQ-C30

SECONDARY OUTCOMES:
Global health-related quality of life | 60 and 90 days
Pleurodesis failure rate | 30, 60 and 90 days
  Subsequent pleural intervention required on same side as pleurodesis
  Chest X-ray opacification greater than 25% on side of intervention
Improvement in symptoms of pain and breathlessness | 30, 60 and 90 days
  Medical Research Council (MRC) dyspnoea scale 100mm Visual Analog Scale for pain and breathlessness
Complication rate | Day 7, 14, 30, 60 and 90
  Clinical review and adverse event documentation

CONTACTS AND LOCATIONS:
Locations (1):
- Guy's and St Thomas' NHS Foundation Trust, London, United Kingdom